CLINICAL TRIAL: NCT00932490
Title: Tailored Intervention Protocol for Oral Chemotherapy Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00015563; 1R15CA139398-01 (NIH); 3031779
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2012-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse Coaching (Experimental): Tailored adherence intervention that will be based on the particular needs of patients and an advanced practice nurse will suggest individualized strategies to overcome barriers to adherence
  Interventions: Behavioral: Nurse Coaching
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Nurse Coaching — Tailored adherence intervention that will be based on the particular needs of patients and advanced practice nurses will suggest individualized strategies to overcome barriers to adherence
  Arms: Nurse Coaching

SUMMARY:
The primary aim of study is to:

1. Test the effectiveness of a tailored protocol in promoting adherence to oral chemotherapeutic agents in adults receiving a new oral chemotherapeutic agent for breast, colorectal, GIST, renal cell,and hepatocellular cancers.

   Exploratory Aims:
2. Examine adherence to oral chemotherapeutic agents over time at 2, 4 and 6 months in a sample of breast, colorectal, GIST, renal cell,and HPCC cancers patients.
3. Examine the effects of age, gender, caregiver availability, personal involvement in health care, and depression on adherence to oral chemotherapeutic agents.

DETAILED DESCRIPTION:
While cancer patients express a preference for oral medications, compliance to these medications varies. Patients who successfully adhere to chemotherapy regimens have a greater chance of non-recurrence and long-term quality of life. Thus, helping patients tolerate oral chemotherapy regimens is critical to their survival. The aims of this study are to 1) test the effectiveness of a tailored protocol to promote adherence to oral chemotherapeutic agents in adults receiving treatment for cancer, 2) examine adherence to oral chemotherapeutic agents over time, and 3) examine the effects of age, gender, caregiver availability, personal involvement in health care, and depression on adherence rates to oral chemotherapeutic agents.

The tailored adherence protocol is based on the self-regulatory model of adherence. The intervention identifies patient knowledge, behavioral skills, and affective support and tailors adherence strategies or overcomes barriers in each of these three categories. A randomized clinical trial will examine the adherence rates in a 150 adults started on a new oral chemotherapeutic agent. A control group will receive standard chemotherapy education. Participants in the experimental group will receive the standard education, an assessment and the tailored intervention developed by an advanced practice nurse. The intervention will be administered via telephone calls over six months. Patient adherence rates will be measured in both groups at 2, 4 and 6 months using self report, symptom profiles, and pharmacy fill rates. To determine the effectiveness of the adherence protocol, we will use Generalized Estimating Equations (with SAS), which provide a unified approach to longitudinal modeling techniques for normally and non-normally distributed outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of Breast, Colorectal, GIST, Renal, HPCC, Myeloma and Chronic Leukemia
* 18 years or older
* a treatment regimen that includes at least one oral chemotherapeutic agent
* ability to read and write English
* ability to give informed consent
* ability to have prescriptions for oral chemotherapy filled at the Duke University Medical Center pharmacy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Adherence to Oral Chemotherapy Medication | 2, 4, & 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Susan M Schneider, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Schneider SM, Hess K, Gosselin T. Interventions to promote adherence with oral agents. Semin Oncol Nurs. 2011 May;27(2):133-41. doi: 10.1016/j.soncn.2011.02.005. PMID 21514482